CLINICAL TRIAL: NCT01438554
Title: Phase I Study Determining the Safety and Tolerability of Combination Therapy With Pazopanib, a VEGFR/PDGFR/Raf Inhibitor, and GSK1120212, a MEK Inhibitor, in Advanced Solid Tumors Enriched With Patients With Advanced Differentiated Thyroid Cancer, Soft Tissue Sarcoma, and Cholangiocarcinoma
Brief Title: Phase 1 Study of Pazopanib With GSK1120212 in Advanced Solid Tumors, Enriched With Patients With Differentiated Thyroid Cancer, Soft-tissue Sarcoma, and Cholangiocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Comprehensive Cancer Network (Network); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J1162; NA_00048646 (Other: JHMIRB)
Record Dates: First submitted 2011-08-23; First posted 2011-09-22 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Solid Tumors; Thyroid Cancer; Soft-tissue Sarcoma; Cholangiocarcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Sarcoma; Cholangiocarcinoma | interventions — pazopanib; trametinib

ARMS (1):
- Pazopanib and GSK1120212 (Experimental): Treatment will be administered on an outpatient basis. Both drugs are taken orally. Each cycle lasts 28 days. The doses of each drug will depend on when patient enters study.
  Interventions: Drug: Pazopanib; Drug: GSK1120212

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient
Drug: GSK1120212
  Other Names: Trametinib; Mekinist

SUMMARY:
The purpose of this study is to determine the safety and toxicity of the combination of pazopanib and GSK1120212 in patients with solid tumors and identify the maximum tolerated dose (MTD) of this combination for phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation cohort for all solid tumors is closed to enrollment.
* Expansion cohorts: Soft-tissue sarcoma, cholangiocarcinoma, and differentiated thyroid cancer (DTC) cohorts are closed to enrollment. Patients in the DTC cohort must have disease that is able to be biopsied.
* Must have measurable disease.
* Tumor progression in the 6-month period prior to study drug initiation.
* DTC patients: must have radioiodine non-avid lesions, OR radioiodine avid lesions that have not responded to treatment with radioactive iodine.
* ECOG performance status less than or equal to 1.
* Life expectancy >3 months.
* Blood pressure <140 mmHg and <90 mmHg.
* LVEF is >= 50%
* Must be able to swallow pills.

Exclusion Criteria:

* Chemotherapy, radiotherapy, other investigational therapy, or major surgery within 4 weeks.
* Sarcoma and cholangiocarcinoma ONLY: Prior VEGF-targeted TKI therapy.
* Pregnant or currently breastfeeding.
* Unresolved toxicity greater than grade 1.
* Evidence of active hepatitis or HIV.
* Significant cardiovascular disease.
* Taking medications known to be strong inducers or inhibitors of CYP3A enzymes.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
* History of gastrointestinal condition causing malabsorption or obstruction.
* Cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep vein thrombosis (DVT) within past 6 months.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase risk of pulmonary hemorrhage.
* Hemoptysis within 6 months of starting treatment.
* History of retinal vein occlusion (RVO) or central serous retinopathy (CSR), or predisposing factors to RVO or CSR as assessed by ophthalmic exam.
* Known brain mets that are not stable for at least 8 weeks prior to treatment, or patient is on glucocorticoids for brain mets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of pazopanib and GSK1120212 when combined in patients with solid tumors | Approximately one year
Adverse events as a measure of the safety and tolerability profile of pazopanib in combination with GSK1120212 in patients with solid tumors | Approximately two years

SECONDARY OUTCOMES:
Objective response rate at six months in patients with advanced thyroid cancer, soft tissue sarcoma and cholangiocarcinoma being treated at the MTD | Approximately one year
Progression-free survival (PFS) in patients with advanced thyroid cancer, soft tissue sarcoma and cholangiocarcinoma being treated at MTD. | Approximately one year
Correlation of PK data with radiographic response, PD markers, and the impact of tumor histologic subtype and tumor genotype on radiographic response for patients with advanced thyroid cancer | Approximately one year
PD marker analysis on peripheral blood mononuclear cells for patients with soft tissue sarcoma and cholangiocarcinoma | Approximately one year

CONTACTS AND LOCATIONS:
Overall Officials: Nilo Azad, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - MD Anderson Cancer Center, Houston, Texas